CLINICAL TRIAL: NCT04027231
Title: Comportement Electrochimique D'alliages Biomedicaux Dans Des Liquides Synoviaux En Fonction De L'etat Pathologique
Brief Title: Electrochemical Behavior of Biomedical Alloys Exposed to Human Synovial Fluid
Status: Completed | Type: Observational
Sponsor: Brigitte Jolles, MD (Other)
Responsible Party: Sponsor-Investigator, Brigitte Jolles, MD, Professor, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Other Study IDs: 208/13
Record Dates: First submitted 2019-05-24; First posted 2019-07-19 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-12

CONDITIONS: Arthroplasty, Replacement, Knee; Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Ahlback I
  Interventions: Other: analysis of the synovial fluid
- Ahlback II
  Interventions: Other: analysis of the synovial fluid
- Ahlback III
  Interventions: Other: analysis of the synovial fluid
- 1 year following TKA
  Interventions: Other: analysis of the synovial fluid
- TKA revision
  Interventions: Other: analysis of the synovial fluid

INTERVENTIONS:
Other: analysis of the synovial fluid — Electrochemical cell analysing the patients' synovial fluid whenever an invasive intervention is medically prescribed

SUMMARY:
Biomedical implant metals are reactive when in contact with body fluids. Some reactions may adverse the biocompatibility character of the material and should be studied. This can be achieved by direct measurement through electrochemical, gravimetric, spectrophotometric and surface analysis of reaction occurring at the interface between functionalized metal samples and body fluids (synovia) directly extracted from patients.

The general aim of this project is to contribute to develop a comprehensive vision of interfacial reactions occurring on biomedical alloy surfaces exposed to human synovial fluid and to link them to clinical data

DETAILED DESCRIPTION:
Most widely used biomedical materials are polymeric, ceramics and metals. Among these materials, metals exhibit a unique combination of mechanical strength, toughness, wear resistance and forming easiness. Metals are chemically reactive when in contact with body fluids. While some of the reactions are welcome, such as the surface oxidation providing corrosion protection, other reactions may adverse the biocompatibility character of the material.The understanding of these reactions is the object of several studies. Corrosion scientists try to characterise the corrosion response of metals when in contact with simulated body fluids in order to verify the occurrence of hypothetical mechanisms. Biologists look at specific reaction products expected to be released by cells when set in contact with structured or functionalized surfaces. These approaches are necessary but also time consuming due to the complexity of possible reaction mechanisms. As complement to these deductive approaches we propose here an inductive one based on direct measurement through electrochemical, gravimetric, spectrophotometric and surface analysis of reaction occurring at the interface between functionalized metal samples and body fluids (synovia) directly extracted from patients.

The general aim of this project is to contribute to develop a comprehensive vision of interfacial reactions occurring on biomedical alloy surfaces exposed to human synovial fluid and to link them to clinical data. This will be achieved through a collaboration between surgeons and corrosion scientists. The synovial fluid will be extracted form patients using an established procedure and transferred to a portable sterile corrosion laboratory located close to the surgery room. There, surface reaction will be characterized using electrochemical methods already successfully applied in recent studies carried out by the same team. We will be integrating in-situ quartz crystal microgravimetry and in-situ Raman spectroscopy as well as ex-situ methods. Further, metal surfaces will be chemically functionalized (wettability, oxidation, surface charge) in order to selectively influence specific reactions of body fluid components (i.e. adsorption depends on surface energy and wettability while Redox reactions are influenced by the oxidation state of the surface. The acquired information will be compared to the clinical state of the patient in order to establish possible correlations between interface reactivity and patient state.

ELIGIBILITY:
Inclusion Criteria:

* indication to knee joint puncture
* Written consent

Exclusion Criteria:

* refusing to sign written consent
* patient unabled to have a follow-up by their own surgeon/doctor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Human adults presenting either a knee osteoarthritis, a knee joint replacement at 1-year follow-up or an indication for TKA revision surgery
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Open circuit potential | only 1 measurement immediatly after collection, the day of collection (1 day)
  through a potentiostat device
Changes in Corrosion speed | only 1 serie of measurements immediatly after collection, every 10 minutes, during 1 day
  through polarisation resistance
Changes in electrochemical impedance spectrum | only one serie of measurements after collection, every 60 minutes, during 1 day
  through electrochemical impedance spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV - Site HO, Lausanne, CH, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided